CLINICAL TRIAL: NCT04146532
Title: Effects of Aspirin on Emotional Reactivity, Memory, and Risk-taking
Brief Title: Aspirin Effects on Emotional Reactions
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Baldwin Way, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2019H0262
Record Dates: First submitted 2019-10-28; First posted 2019-10-31 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Healthy Adults
Keywords: Aspirin; Acetylsalicylic acid; Emotional reactivity; Memory; Risk-taking; Inflammation
MeSH Terms: conditions — Risk-Taking; Inflammation | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Note. 135 of an originally intended 200 participants had been enrolled at the time of cessation of research activities due to COVID-19 research closures. Therefore, the intended sample was increased to 270 to allow comparison between pre-COVID and post-COVID participants.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Single dose of a 500mg placebo tablet.
  Interventions: Drug: Placebo
- Aspirin 500MG (Active Comparator): Single dose of a 500 mg aspirin tablet.
  Interventions: Drug: Aspirin 500 MG

INTERVENTIONS:
Drug: Aspirin 500 MG — Single 500mg aspirin capsule.
  Other Names: actelysalicylic acid
  Arms: Aspirin 500MG
Drug: Placebo — Single 500mg placebo capsule.
  Arms: Placebo

SUMMARY:
The aim of this study is to determine whether the drug aspirin has effects on emotional reactivity, emotional memory, and risk-taking behaviors.

DETAILED DESCRIPTION:
The goal of this study is to determine if aspirin (acetylsalicylic acid) alters emotional reactions to emotion evoking pictures as well as memory for them. Using a double-blind parallel arm study, participants will receive either placebo or a pain-relieving dose of aspirin (500mg). One hour later they will complete 30 minutes of tasks. This will include ratings of emotional pictures and memory for them. The paradigm is similar to previous experiments done in this lab using other cyclooxygenase inhibitors: ibuprofen and acetaminophen (Durso, Luttrell, & Way, 2015; Psychological Science, https://doi.org/10.1177/0956797615570366). Risk taking on the Balloon Analogue Risk Task will also be assessed. Participants will be healthy young adult males at Ohio State University.

ELIGIBILITY:
Inclusion Criteria:

At least 18 years old and biologically male

Exclusion Criteria:

Due to the use of aspirin in this study, women will be excluded from the study due to potential negative effects it may have on pregnancy

Participants will also be excluded for the following medical reasons:

1. Having an allergy to aspirin, other salicylates, or any other pain reliever/fever reducer.
2. Having or recovering from a viral infection such as the chicken pox or flu.
3. Having taken aspirin or another NSAID drug (aspirin, ibuprofen, naproxen, or others) within the last 8 hours or plan to take aspirin or another NSAID drug in the 8 hours after the end of the study.
4. Having more than three drinks of alcohol in the 8 hours after completion of the study.
5. Having asthma, hay fever, nasal polyps, or chronic respiratory disease.
6. Impaired liver/kidney or impaired cardiovascular circulation (renal vascular disease, congestive heart failure, volume depletion, major surgery, sepsis or major hemorrhagic events)
7. Active or severe liver or kidney disease.
8. An ulcer, history of ulcers or are prone to bleeding.
9. A history of blood clotting defects.
10. Severe anemia.
11. Taking any of the following drugs: A blood thinning anticoagulant (e.g. warfarin), Digoxin, An Angiotensin Converting Enzyme (ACE) Inhibitor, Methotrexate, An oral glucocorticoid (e.g. hydrocortisone),Valproic Acid, A Selective Serotonin Reuptake Inhibitor (SSRI; e.g. Prozac; Zoloft)
12. Have had stomach ulcers or bleeding problems.
13. Have stomach problems such as heartburn, upset stomach, or stomach pain that does not go away or reoccurs.
14. Surgery in the last week or will have a surgery in the next week.
15. High blood pressure.
16. Diabetes, gout, or arthritis.
17. Low uric acid or Glucose-6-phosphate dehydrogenase (G6PD) deficiency.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be biologically male to participate in study.
Enrollment: 268 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Emotional Reactivity | 1.5 hours
  Changes in self-reported evaluations of valence on a 1 to 7 scale and felt reactions to emotional images on a 1-7 scale.
Memory | 1.5 hours
  Changes in memory for emotional pictures. After rating the images, the participants will be shown them again as well as new pictures and asked to indicate whether they have seen the picture before or not.
Risk-Taking | 1.5 hours
  We will measure the adjusted average number of pumps on the Balloon Analogue Risk Task.

SECONDARY OUTCOMES:
Individual Differences | 1.5 hours
  Self-reported political ideology will be examined as a moderator of the self-reported ratings of the images as well as memory for them.

CONTACTS AND LOCATIONS:
Locations (1):
- Psychology Building, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made available online for responses to the tasks.
Supporting Information: Study Protocol, SAP
Time Frame: The dataset and annotation will be made available by 7/1/2023

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT04146532/Prot_SAP_000.pdf